CLINICAL TRIAL: NCT07400913
Title: Implementation of Long-read Sequencing for Epimutation Detection in the Diagnosis of Rare Diseases.
Brief Title: Implementation of Long-read Sequencing for the Diagnosis of Rare Diseases.
Acronym: LongEpi
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2025/103
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Rare Diseases; Albinism; Intellectual Disability
Keywords: Rare diseases; Long-read sequencing; Epimutation
MeSH Terms: conditions — Rare Diseases; Albinism; Intellectual Disability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — DNA
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients
  Interventions: Genetic: Long-read sequencing

INTERVENTIONS:
Genetic: Long-read sequencing — Long-read sequencing

SUMMARY:
Following on from the third national plan for rare diseases (PNMR3), the main objectives of the PNMR4 are to reduce diagnostic uncertainty and dead ends and to strengthen translational research to promote diagnosis and the development of new treatments in the field of rare diseases.

To this end, the French Genomic Medicine Plan 2025 (PFMG2025) is organizing the rollout of whole genome sequencing (WGS) for diagnostic purposes.

This technological milestone, covering regions outside the coding regions, has recently enabled the identification of variations in the RNU4-2 gene as a major cause of Intellectual Developmental Disorder (IDD), accounting for approximately 0.4% of cases. RNU4-2 is a gene encoding a small nuclear RNA (snRNA), which is not translated into protein, and whose variations are not accessible to exome sequencing techniques.

However, based on current knowledge, these techniques are based on short-read sequencing technology and can diagnose up to 50% of patients. It is therefore necessary to develop new techniques to detect variations not identified by these techniques.

In this context, the development of third-generation sequencing, particularly using Nanopore technology, now makes it possible to combine genomic and post-genomic approaches through long-read whole genome sequencing coupled with the detection of methylated cytosines on native DNA.

This new approach therefore enables the simultaneous detection of point or structural genomic variants, methylation abnormalities, and haplotype reconstruction. Numerous studies have shown that this strategy improves the diagnosis rate of rare diseases and could become a first-line genetic test.

DNA methylation is an epigenetic modification that does not cause changes in the genomic sequence but regulates the transcription (RNA synthesis) of genes and therefore their expression. Methylation studies are performed either to establish an episignature or to search for methylation abnormalities. An episignature is the result of a variation in a gene known to regulate methylation marks.

Methylation abnormalities are already known and sought after in targeted analysis for certain diseases such as Prader-Willi/Angelman syndromes and Beckwith-Wiedemann/Silver-Russell syndromes. The contribution of methylation analysis to the diagnosis of other diseases has recently been demonstrated. For example, in methylmalonic aciduria and homocystinuria type cblC associated with the autosomal recessive gene MMACHC, promoter methylation analysis revealed hypermethylation linked to the presence of an intronic variant of the PRDX1 gene. This intronic variant leads to the synthesis of an aberrant antisense RNA overlapping the promoter of the MMACHC gene, causing its hypermethylation. In 2024, combined whole-genome and methylation analysis in patients with porokeratosis led to the discovery of the FDFT1 gene. In general, the study of methylation profiles has shown its value in reducing diagnostic uncertainty in patients with rare diseases who have not been diagnosed after genome analysis.

The search for methylation abnormalities (or epimutation) at the pan-genomic level in the context of molecular diagnosis of rare diseases remains largely inaccessible and poorly described in the literature. The techniques routinely used for their detection are most often based on bisulfite treatment and PCR amplification. The disadvantages of bisulfite treatment are that it degrades DNA, preventing long-read applications, that it does not distinguish between 5mC and 5hmC methylation, and that failure to treat unmethylated cytosines can lead to false positives . In addition, phase determination with a genomic variant identified in short reads requires complementary techniques such as SNP arrays.

This approach therefore appears to be a major technological advance in the fight against diagnostic uncertainty in rare diseases and is part of the move towards precision medicine for patients.

As part of our Reference Center for Developmental Anomalies and Malformation Syndromes of Southwest Occitanie Réunion (CRMR ADSOOR) at Bordeaux University Hospital, we have developed clinical and molecular expertise, particularly in the field of developmental anomalies with intellectual development disorders (particularly chromatinopathies and Rubinstein Taybi syndrome and albinism.

In 2024, 2,300 consultations were carried out at the CRMR. In addition, 243 and 228 genome or exome analyses were interpreted in our molecular biology laboratory for albinism and intellectual development disorder and malformation syndrome, respectively.

Our expertise in these two areas therefore represents the best starting point for the development of this pilot project using this innovative approach at Bordeaux University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients,adults under guardianship, or minors with autorisation from their legal representative, for whom extracted DNA or a tube of frozen blood is available in the molecular genetics laboratory.
* Patients investigated for either :

  * a syndromic intellectual development disorder (IDD) defined by:
* age :

  * Between 0 and 5 years with strict criteria: severe developmental delay in terms of motor skills, language and/or sociability OR
  * ≥ 6 years: patients with IDD, regardless of severity (but with IDD proven by ad hoc neuropsychological tests)
* association with minor morphological criteria and/or organ malformations.

  * albinism defined by the presence of two of the following clinical signs: foveal hypoplasia, retinal hypopigmentation, iris transillumination, crossed asymmetry, nystagmus, skin/hair hypopigmentation (suggested diagnostic criteria proposed by Kruitj et al. (PMID: 30098354)).
* Patients for whom genetic analyses (panel, exome, genome) are either :

  * inconclusive (no pathogenic or probably pathogenic variant).
  * A single heterozygous pathogenic or probably pathogenic variant identified in a gene associated with an autosomal recessive disease compatible with the phenotype.

Exclusion Criteria:

* Refusal to participate in research protocols expressed at the time of written consent for genetic analysis as part of medical care.
* Opposition expressed following receipt of information note.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients for whom extracted DNA or a tube of frozen blood is available in the molecular genetics laboratory and for which genetic analysis were unconclusive.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Methylation anomalies | Baseline
  Detection of hypermethylated CpG islets in a locus close to a gene known in human pathology and associated with a phenotype compatible with the patient's clinical presentation

CONTACTS AND LOCATIONS:
Overall Officials: Julien VAN-GILS, MD, Principal Investigator — CHU Bordeaux - Hôpital Pellegrin
Locations (1):
- CHU Bordeaux - Hôpital Pellegrin, Bordeaux, France